CLINICAL TRIAL: NCT02988843
Title: Phase II Study of Brentuximab Vedotin and Bevacizumab in Men With Refractory CD-30 Positive Germ Cell Tumors
Brief Title: Study of Brentuximab Vedotin And Bevacizumab In Refractory CD-30 Positive Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding Unavailable
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS190
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Germ Cell Tumor
Keywords: GCT
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Brentuximab Vedotin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin & Bevacizumab (Experimental): * Bevacizumab will be administered at a dose of 15 mg/kg IV every 21 days; over 90 minutes during 1st infusion, over 60 minutes as 2nd infusion and over 30 minutes for subsequent infusions if prior infusions well tolerated.
  * Brentuximab vedotin will be administered first at 1.8 mg/kg (maximum dose of 180 mg) IV over 30 minutes every 21 days.
  Interventions: Drug: Brentuximab Vedotin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Dose level 1: 1.8 mg/kg every 21 days (up to 180 mg) Dose level -1 :1.2 mg/kg every 21 days ( up to 120 mg)
  Other Names: ADCETRIS
Drug: Bevacizumab — 15 mg/kg every 21 days
  Other Names: Avastin

SUMMARY:
This is a multi-center phase II study of brentuximab vedotin in combination with bevacizumab for the treatment of refractory CD-30+ germ cell tumors (GCT) after disease progression on imaging and/or tumor marker progression documented by serially rising alpha-fetoprotein (AFP) or beta human chorionic gonadotropin (bHCG) measured on at least 2 consecutive visits and determined by treating physician to be clinically significant. Patients unable to receive 2nd line of platinum-based chemotherapy due to toxicity or refusal would also be eligible.

ELIGIBILITY:
Inclusion Criteria:

* Male, ≥ 18 years of age
* Diagnosis of CD-30 positive germ cell tumor. CD30 expression will be tested by immunohistochemistry (IHC) in archival or fresh tumor tissue as is routinely done for diagnosis.
* Disease progression on imaging or tumor marker progression (clinical significance of tumor marker progression to be decided per the discretion of treating physician) after at least 2 lines of platinum-based chemotherapies unless patient is ineligible for further platinum based chemotherapy or refuses 2nd line platinum based chemotherapy due to toxicity. For primary mediastinal germ cell tumors, failure of first-line chemotherapy will be accepted. Prior high dose chemotherapy with hematopoietic stem cell rescue is allowed. Prior treatment with bevacizumab is allowed.
* At least 3 weeks should have elapsed since the last treatment (e.g. chemotherapy, targeted small molecule therapy, immunotherapy or radiation) and must have recovered to grade 1 or better from the acute effects of prior therapy.
* Presence of measurable disease according to RECIST 1.1
* ECOG performance status 0 or 1
* Adequate marrow and organ function within 28 days prior to study registration as defined below:

  * Leukocytes > 3,000/µL
  * ANC > 1500/µL
  * Hemoglobin ≥ 9 g/dL, Note: Blood transfusion will be allowed for patients with hemoglobin < 9 g/dl and G-CSF is allowed for neutropenic patients at time of enrollment.
  * Platelets > 100,000/mm3
  * Creatinine: ≤3mg/dl OR if serum creatinine > 3 mg/dl, estimated GFR >30 mL/min/1.73m2
  * INR: <1.5 x institutional upper limit of normal OR < 3 if on warfarin or other anticoagulants. There should be no evidence of active bleeding while on anticoagulants.
  * Total bilirubin: ≤ 2 x institutional upper limit of normal (ULN)
  * SGOT (AST) or SGPT (ALT): < 3 x institutional upper limit of normal (< 5 x ULN if liver metastases present)
  * Proteinuria: If patient has proteinuria, it should be <2+ (< 100 mg/dl or per institutional guidelines). If proteinuria is 2+ or greater (≥ 100 mg/dl per institutional guidelines), patients should undergo a 24- hour urine collection and 24 hour urinary protein should be less than < 2 grams.
* Sexually active men with partners of women of childbearing potential must agree to practice effective methods of contraception during the study and for 6 months after the last treatment
* Provide voluntary written consent and HIPAA authorization for release of personal health information, approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC)

Exclusion Criteria:

* Prior treatment with Brentuximab Vedotin.
* Known active brain metastases and or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided brain metastases are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study registration. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* History of blood clots, pulmonary embolism, or deep vein thrombosis in previous 6 months unless controlled by anticoagulant treatment
* Known history of HIV
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Received a live vaccine within 1 week prior to the first dose of study treatment
* Has active autoimmune disease that required systemic treatment with use of disease modifying agents, corticosteroids or immunosuppressive drugs
* Any clinically significant active infection that requires systemic treatment at the time of enrollment.
* Known allergy to bevacizumab or brentuximab vedotin or any of its excipients
* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction (MI) within 6 months of study registration
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess in previous 6 months
* Prior major surgery within the previous 28 days of study registration and/or presence of any non-healing wound, fracture, or ulcer.
* Use of an investigational agent within the previous 28 days of study registration.
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥150 mmHg and/or diastolic blood pressure (DBP) of ≥ 90mmHg]. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study registration
* Arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or MI within 6 months of study registration
* History of posterior reversible encephalopathy syndrome
* Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy > than 6 months prior to study entry
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Concurrent use of rifampin or ketoconazole

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Gupta, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Brentuximab Vedotin & Bevacizumab: * Bevacizumab will be administered at a dose of 15 mg/kg IV every 21 days; over 90 minutes during 1st infusion, over 60 minutes as 2nd infusion and over 30 minutes for subsequent infusions if prior infusions well tolerated.
  * Brentuximab vedotin will be administered first at 1.8 mg/kg (maximum dose of 180 mg) IV over 30 minutes every 21 days.
  Brentuximab Vedotin: Dose level 1: 1.8 mg/kg every 21 days (up to 180 mg) Dose level -1 :1.2 mg/kg every 21 days ( up to 120 mg)
  Bevacizumab: 15 mg/kg every 21 days
Period: Overall Study
Arm/Group | Brentuximab Vedotin & Bevacizumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Brentuximab Vedotin & Bevacizumab: Bevacizumab will be administered at a dose of 15 mg/kg IV every 21 days; over 90 minutes during 1st infusion, over 60 minutes as 2nd infusion and over 30 minutes for subsequent infusions if prior infusions well tolerated. Brentuximab vedotin will be administered first at 1.8 mg/kg (maximum dose of 180 mg) IV over 30 minutes every 21 days
Arm/Group | Brentuximab Vedotin & Bevacizumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Response Rate as Defined by the RECIST 1.1 Criteria, Integrated With Tumor Marker Response.
Description: Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
  In addition to CT scan to assess for disease evaluation, whole body bone scans will be done for patients with known or suspected bone metastases to assess for bone lesions.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin & Bevacizumab
Number analyzed (Participants) | 1
Participants
  Baseline | 1
  Complete Remission | 0
  Progressive disease | 0

2. Secondary Outcome: Number of Participants Experiencing Progression Free Survival
Description: Incidence of Progression-free survival - Number of patients who were alive and did not have disease progression
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin & Bevacizumab
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Number of Participants Who Were Alive at 2 Years - Overall Survival
Description: Number of participants who were alive at 2 years (Overall survival)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin & Bevacizumab
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE) and Severe Adverse Events (SAE)
Description: Safety/ toxicity of brentuximab vedotin, measured by incidence of AEs/SAEs
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin & Bevacizumab
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Brentuximab Vedotin & Bevacizumab
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin & Bevacizumab (N=1)
Chills (General disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT02988843/Prot_SAP_000.pdf